CLINICAL TRIAL: NCT03212027
Title: Preoperative Prediction of the Pathological Classification of Thymic Epithelial Tumors by Apparent Diffusion Coefficient Using Ultra-high B-values
Brief Title: Preoperative Prediction of of Thymic Epithelial Tumors by Diffusion-Weighted MR Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016SF-211
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Thymic Epithelial Tumor
Keywords: apparent diffusion coefficient; aquaporins
MeSH Terms: conditions — Thymic epithelial tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with low-risk thymomas: low-risk thymomas include types A, AB, and B1 thymomas
- Patients with high-risk thymomas: high-risk thymomas include types B2 and B3 thymomas
- Patients with thymic carcinomas: thymic carcinomas also called types C thymomas

SUMMARY:
The aim of this study is to analyze aquaporins expression of thymic epithelial tumors and to compare them with apparent diffusion coefficient(ADC) from ultra-high b-values, and to test a possibility of use of ADCuh to identify the pathological type of tumor.

DETAILED DESCRIPTION:
Magnetic resonance (MR) diffusion-weighted imaging (DWI) measures water diffusion in biological tissue. The quantification of diffusion is described by the apparent diffusion coefficient (ADC),which largely depends on the number and separation of barriers.Thus, ADC can provide information regarding tissue microstructure.

According to the literature, ADC is also related to cell membrane permeability for water molecules.It is well known that cellular water transport depends on aquaporins (AQPs).In general,the expression of aquaporins might differ in several pathologic disorders. With reference to this fact,we hypothesize that AQPs expression may influence ADC in thymic epithelial tumors(TETs).Therefore,the aim of the present study is to analyze possible associations between ADC from ultra-high b-values and AQPs expression(ADCuh) in TETs and to use ADCuh to identify the pathological type of tumor.

ELIGIBILITY:
Inclusion Criteria:

* no use of corticosteroid drugs;
* no MRI contraindication;
* no infection or fever;
* tumor diameter is greater than 2cm.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thymic epithelial tumors
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-07-31 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Different DWI parameters in thymic epithelial tumors | 6 months

SECONDARY OUTCOMES:
To acquire aquaporins expression level of thymic epithelial tumors | 6 months